CLINICAL TRIAL: NCT02948036
Title: A Closed-loop Assessment and Treatment Platform for Unipolar Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-1011-16; 1R43MH111325 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-10-28 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 2-methylcyclopentadienyl manganese tricarbonyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MMT (Experimental): Mobile-device, plasticity-based adaptive cognitive treatment
  Interventions: Other: Mobile-device, plasticity-based adaptive cognitive treatment

INTERVENTIONS:
Other: Mobile-device, plasticity-based adaptive cognitive treatment — This study employs a mobile-device delivered treatment program. Participants will be asked to use the assigned treatment program for approximately 30 minutes per session, up to seven sessions per week, over 6 weeks (42 total sessions).
  Other Names: MMT

SUMMARY:
Specific Aim 1: Finalize development of the closed-loop strategy in the MMT application.

Specific Aim 2: Evaluate the acceptability and feasibility of the MMT application with the target population to prepare for a large-scale efficacy trial.

DETAILED DESCRIPTION:
Specific Aim 1: Investigators have recently constructed a beta version of the MMT application, comprised of the multi-modal assessment modules, several treatment modules and an initial version of the closed-loop algorithm to control treatment delivery. Utilizing the extensive experience in developing mobile assessment and treatment tools at Posit Science Corporation, the investigators will employ an iterative development process incorporating feedback from users (focus groups of patients with mood disorders), clinicians and scientists (project consultants) to achieve the following development goals: (1) Finalize MMT's closed-loop algorithm to incorporate all assessment modules and expand the existing triage approach; (2) Expand cognitive behavioral therapy (CBT) functions within the app; and (3) Expand in-app bi-directional communication feature between the clinician and user. At the completion of Specific Aim 1, the investigators will have a mobile app suitable for evaluation in a feasibility trial (Specific Aim 2).

Specific Aim 2: The investigators will conduct a single arm, open label feasibility field trial with 40 participants that meet criteria for Major Depressive Disorder (MDD). Participants will be asked to engage with the experimental cognitive treatment and spend up to six weeks engaged in 15 hours of cognitive training as an adjunct to their standard clinical treatment. The experimental cognitive treatment will be deployed as dictated by the closed loop predictive algorithm, with all patient data continuously accessible for remote monitoring by the attending clinicians, research staff and Principal Investigator at University of Minnesota, and research staff and Sponsor PI at Posit Science Corporation. Participants will be re-evaluated every two weeks during treatment use, and again at the expected time of completion of training, at 6 weeks, to evaluate changes in cognitive function. Participants will then stop using their assigned program for 6 weeks, and return for a follow-up assessment to evaluate the endurance of changes in cognitive function in the absence of further program use.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 60 years of age.
2. Participant must score ≥ 9 on the Patient Health Questionnaire-9 (PHQ-9).
3. Participant taking antidepressants or engaged in psychotherapy will not be excluded. If potential participants are currently prescribed psychotropic medication, they must be on a clinically stable medication regimen for ≥ 6 weeks prior to screening, based on self-report or as verified by medical health records, when available and authorized.
4. Participant must be a fluent English speaker.
5. Participant must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control and use a mobile device and/or computer as required to complete study activities.
6. Participant must have access to wireless Internet connectivity.
7. Participant must be willing to communicate with study staff via email.

Exclusion Criteria:

1. Participant with unstable and/or untreated conditions that may affect cognition, including untreated substance abuse/dependence disorders, unmanaged cardiovascular disease, endocrine or neurologic disorder, epilepsy, brain injury, hospitalization within 6-weeks of enrollment, ongoing chemotherapy or other cancer treatment (e.g., radiation) .
2. Participant with history or current DSM-5 diagnosis of psychosis, such as schizophrenia, schizoaffective disorder, delusion disorder, psychotic disorder NOS, bipolar disorder, substance abuse (<1 year), and/or mood congruent or mood incongruent psychotic features or disorders.
3. Participant has a history or current diagnosis of dementia and/or scores less than a 14 (75%) on the UBACC.
4. Participant with active suicidal ideations or behaviors within 2 months of screening.
5. Participant that shows signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) during any in person visit. Such participants will have that visit re-scheduled; participants with this problem occurring more than once may be excluded and dropped at the discretion of the Principal Investigators.
6. Participant has problems performing assessments or comprehending or following spoken instructions, or those with behaviors during screening or baseline visits that, in the judgment of the screening staff, are likely to present significant problems for the staff conducting assessments.
7. Participant is enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment that could affect the outcome of this study. However, participation in standard treatments (e.g., occupational therapy) or use of prescribed medications (e.g., anti-depressants) is allowable..
8. Participant is using computer-based cognitive training programs or has used it within a month of the consent date.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Change in total score for depressive symptoms using Beck Depression Scale (BDI-II) | At 2 weeks, 4 weeks, 6 weeks and at 12 weeks
  The Beck Depression Scale (BDI-II) is a self-report questionnaire that assesses depressive symptoms with a scoring range between 0-63.

SECONDARY OUTCOMES:
Change in total score for depressive symptoms using Patient Health Questionnaire (PHQ-9) | At 2 weeks, 4 weeks, 6 weeks and at 12 weeks
  The Patient Health Questionnaire (PHQ-9) is a self-report questionnaire that assesses the degree of depression severity with a scoring range between 0-27.
Change in total score for anxiety symptoms using Generalized Anxiety Disorder (GAD-7) | At 2 weeks, 4 weeks, 6 weeks and at 12 weeks
  The Generalized Anxiety Disorder (GAD-7) is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder with a scoring range between 0-21.
Change in total score for mood symptoms using Immediate Mood Scaler (IMS) | At 2 weeks, 4 weeks, 6 weeks and at 12 weeks
  The Immediate Mood Scaler (IMS) is a clinical assessment that assesses momentary mood symptoms related to anxiety and depression with a scoring range between 22-181.
Change in total score for quality of life using the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | At 2 weeks, 4 weeks, 6 weeks and at 12 weeks
  The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) assesses the degree of enjoyment and satisfaction experienced in various areas of daily functioning with a scoring range between 0-70.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Balci, MD, Principal Investigator — University of Minnesota - Department of Psychiatry; Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States